CLINICAL TRIAL: NCT04221919
Title: Different β -Blockers in Patients With ST-segment Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Different β -Blockers in STEMI and Primary PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, MD, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR management
Record Dates: First submitted 2020-01-05; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Primary PCI

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carvedilol (Experimental)
  Interventions: Drug: β -Blockers
- Bisoprolol (Experimental)
  Interventions: Drug: β -Blockers
- Metoprolol tartrate (Experimental)
  Interventions: Drug: β -Blockers
- Metoprolol succinate (Experimental)
  Interventions: Drug: β -Blockers

INTERVENTIONS:
Drug: β -Blockers — Target doses of carvedilol, bisoprolol, metoprolol tartrate, or metroprolol succinate

SUMMARY:
Carvedilol, target dose: 50 mg daily; Bisoprolol, target dose: 10 mg daily; Metoprolol tartrate, target dose: 150 mg daily; Metroprolol succinate, target dose: 200 mg daily

DETAILED DESCRIPTION:
The investigators will investigate the efficacy and safety of different β -blockers, as well as heart rate variability, in STEMI patients undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for primary PCI for STEMI involving the LAD within 12 hours of onset of symptoms. STEMI will be defined as typical ECG changes (ST segment elevation ≥2mm in 2 or more precordial leads) associated with acute chest pain or an elevation of cardiac enzymes;
* Age ≥18 years;
* Informed consent from patient or next of kin.

Exclusion Criteria:

* Nonischaemic Cardiomyopathy;
* Cardiac surgery planed in the 6 months;
* Mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation);
* Renal or hepatic failure;
* Malignancy, HIV, or central nervous system disorder;
* Cardiopulmonary resuscitation >15 min and compromised level of consciousness;
* Cardiogenic shock;
* Current participation in any research study involving investigational drugs or devices;
* No written consensus;
* Previous myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in LVEDV from baseline | 1 to 5 years
  The primary outcome of this study will be the change from baseline in left ventricular end diastolic volume (LVEDV) post-PCI.
Major adverse cardiovascular events (MACE) | 1 to 5 years